CLINICAL TRIAL: NCT06388512
Title: Intraoperative MRI Prone Position Support Frame Design Feasibility Study
Brief Title: iMRI Prone Positioning Frame Design Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Continuum Educational Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00160044
Record Dates: First submitted 2024-04-02; First posted 2024-04-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy; Pulmonary Embolism
Keywords: laser interstitial thermal therapy
MeSH Terms: conditions — Epilepsy; Pulmonary Embolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Prototype positioning device (Experimental): The prototype prone positioning device will be used during neurosurgical procedures utilizing intraoperative MRI.
  Interventions: Device: prototype prone positioning device

INTERVENTIONS:
Device: prototype prone positioning device — The prototype prone positioning device will be used during neurosurgical procedures utilizing intraoperative MRI.

SUMMARY:
The goal of this study is to learn if the prototype adjustable prone positioning frame is a feasible design for use during neurosurgical procedures which utilize intraoperative magnetic resonance imaging (iMRI). The main questions it aims to answer are:

* Is the prototype prone positioning device design feasible for use during neurosurgical procedures which utilize intraoperative MRI?
* Does use of the prototype device place the patient at increased risk of complications compared to the standard positioning pads? Researchers will place patients in the prone position on the prototype device during neurosurgical procedures that utilize intraoperative MRI and observe for any problems with the positioning device or complications attributable to the positioning device.

DETAILED DESCRIPTION:
Laser Interstitial Thermal Therapy (LITT) ablations are neurosurgical procedures which are performed for several indications including brain tumors and epilepsy. LITT procedures are performed utilizing intraoperative magnetic resonance imaging (MRI) scans. Some of these procedures must be performed in the prone position and can last 8 hours or longer. Investigators have observed several minor skin breakdown complications as well as a few major thromboembolic complications during these long prone procedures. Investigators hypothesize that the cause of the major thromboembolic complications are a result of compression of the femoral veins by the gel pads used to support the patient in the prone position. Many long spine surgeries are performed in the prone position and fewer episodes of skin pressure wounds are experienced and no major intraoperative thromboembolic complications. The study team hypothesizes that the difference is the way that the spine surgery pads support the hips does not compress the femoral vein, therefore significantly decreasing the risk of developing a thrombus intraoperatively.

The aim of this project is to design a modular, adjustable plastic frame to support the spine surgery Jackson table chest and hip pads. Investigators will produce a prototype of the frame and test it during LITT procedures. The prototype of the frame will be 3D printed using the 3D printer owned by the Department of Neurosurgery. The hypothesis is that supporting the patient in the prone position using similar positioning methods to those used for spine surgeries will reduce the rate of skin pressure injuries and prevent future major thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

Adult patients undergoing prone laser interstitial thermal therapy procedures for epilepsy at the University of Kansas Medical Center (KUMC).

Exclusion Criteria:

* Patients under the age of 18
* Patients who are unable to provide informed consent for participation in the study
* Weight above the safe threshold for the device (weight capacity will be determined through computational stress analysis prior start of the study)
* Patients who do not speak English fluently enough to provide informed consent in English
* Vulnerable populations including prisoners, pregnant women, and KUMC employees/students.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-09-04 (Estimated); Primary Completion 2025-09-04 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
Number of devices that meet functional requirements | During and immediately after each through study completion, an average of 1 year
  The device will be evaluated for meeting its primary function during each use. The primary function is to support the patient in the prone position in the MRI machine during neurosurgical procedures. Whether it fulfills its function will be determined through feedback received from the staff involved in its use which may include nurses, MRI technologists, anesthesia providers, and surgeons. This will be a pass/fail criteria.
Number of devices that are damaged during use | During and immediately after each through study completion, an average of 1 year
  The device will be inspected for physical damage during and after each use. It will be inspected for bending, cracks, mechanical wear, or any other type of damage which could affect the device's safety or ability to serve its primary function. The type and severity of the damage will be recorded after each use and evaluated by the investigators. This will be a pass/fail criteria.

SECONDARY OUTCOMES:
Number of patients with skin complications | Immediately after each procedure
  Each patient's skin will be examined after each procedure to evaluate for pressure injuries related to the prone positioning device. Size and severity of the skin injuries will be documented.
Number of patients with thromboembolic complications | During and after each procedure until the patient is discharged.
  Each patient will be monitored for thromboembolic complications such as deep vein thrombosis or pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kinsman, MD, Principal Investigator — mkinsman2@kumc.edu
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong B, Yoon SH, Park SY, Song S, Youn A, Hwang JG. Cardiac Arrest from Patient Position Change after Spine Surgery on a Jackson Table. Acute Crit Care. 2019 Feb;34(1):86-91. doi: 10.4266/acc.2016.00794. Epub 2017 Feb 20. PMID 31723910
- [Background] Cho JK, Han JH, Park SW, Kim KS. Deep vein thrombosis after spine operation in prone position with subclavian venous catheterization: a case report. Korean J Anesthesiol. 2014 Jul;67(1):61-5. doi: 10.4097/kjae.2014.67.1.61. Epub 2014 Jul 29. PMID 25097742
- [Background] Gebhard CE, Zellweger N, Gebhard C, Hollinger A, Chrobok L, Stahli D, Schonenberger CM, Todorov A, Aschwanden M, Siegemund M. Prone Positioning as a Potential Risk Factor for Deep Vein Thrombosis in COVID-19 Patients: A Hypothesis Generating Observation. J Clin Med. 2021 Dec 25;11(1):103. doi: 10.3390/jcm11010103. PMID 35011843
- [Background] Kanter DS, Mikkola KM, Patel SR, Parker JA, Goldhaber SZ. Thrombolytic therapy for pulmonary embolism. Frequency of intracranial hemorrhage and associated risk factors. Chest. 1997 May;111(5):1241-5. doi: 10.1378/chest.111.5.1241. PMID 9149576